CLINICAL TRIAL: NCT03685175
Title: Effect of Cardiotoxic Anticancer Therapy on the Metabolism of [1-13C]Pyruvate in Cardiac Mitochondria
Brief Title: Using Hyperpolarized [1-13C]Pyruvate to Detect Cardiotoxicity
Acronym: HPCardiotox
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Vlad Zaha, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 072016-058
Record Dates: First submitted 2017-03-11; First posted 2018-09-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Breast Neoplasms
Keywords: Magnetic Resonance Imaging; Doxorubicin
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Formal Study (Experimental): Hyperpolarized 13C-pyruvate, is injected into patients before receiving cardiotoxic therapy and immediately after, for a cardiac MRI scan
  Interventions: Drug: Formal study using hyperpolarized 13C-pyruvate injection
- Feasibility Study (Experimental): Hyperpolarized 13C-pyruvate injection, is given to patients after completing cardiotoxic therapy, and again at 1 to 6 six months after the first cardiac MRI scan
  Interventions: Drug: Feasible study using hyperpolarized 13C-pyruvate injection

INTERVENTIONS:
Drug: Formal study using hyperpolarized 13C-pyruvate injection — Administration at two visits 1) after completion of cardiotoxic therapy and 2) 1 to 6 months after the first time point following medical therapy (SOC)
  Other Names: Cardiac MRI with injection of hyperpolarized 13C-pyruvate
  Arms: Formal Study
Drug: Feasible study using hyperpolarized 13C-pyruvate injection — Administration at two visits: 1) baseline MRI before administration of cardiotoxic therapy and 2) after completion of cardiotoxic therapy
  Other Names: Cardiac MRI with injection of hyperpolarized 13C-pyruvate
  Arms: Feasibility Study

SUMMARY:
The anthracycline doxorubicin, first introduced in the 1960's, continues to be an effectively utilized antineoplastic drug. Even at relatively low cumulative doses there is risk of cardiotoxicity. However, the incidence of subclinical cardiotoxicity is not known, carrying a potential risk for late effects in cancer survivors. Doxorubicin has systemic toxicity that may contribute to cardiac metabolic stress, but the main cardiotoxic mechanism involves cardiac mitochondria. The primary goal of this study is to detect early changes in the mitochondrial metabolism in situ as a marker for subclinical doxorubicin induced cardiotoxicity. The problem of cardiovascular complications following chemotherapy for breast cancer goes far beyond anthracyclines alone. In addition, other agents such as trastuzumab, and pertuzumab and emerging novel therapies may also promote cardiovascular injury. The secondary objective is to test the hypothesis that cardiotoxicity due to other medical anticancer therapies and radiation therapy involving the heart field is associated with a signature of early impaired aerobic cardiac metabolism through pyruvate dehydrogenase.

DETAILED DESCRIPTION:
This is a prospective, single-center study in women and men with breast cancer requiring cardiotoxic therapy. The study will be conducted in parallel to the standard clinical care, at dedicated visits.

In this study patients will undergo a cardiac magnetic resonance (MR) signal detection after injection of hyperpolarized carbon-13 pyruvate. The study will be performed before the course of cardiotoxic therapy, and after completing the treatment.

Patients will be screened prior to enrollment based on study specific inclusion and exclusion criteria and MRI safety criteria.

On the day of the metabolic cardiac MR scan an IV line will be inserted and the participant will receive a bolus of oral glucose. The ingestion of glucose will be required to prepare the state of the heart for metabolic imaging. Following this preparation the participant will undergo a cardiac MR study of about 45 minutes, including carbon-13 dedicated sequences.

A separate dedicated cardiac MRI session may be completed in certain participants.

Feasibility Study (Part I) : Administration at two visits 1) after completion of cardiotoxic therapy and 2) 1 to 6 months after the first time point following medical therapy (SOC).

Formal Study (Part II) : Administration at two visits: 1) baseline MRI before administration of cardiotoxic therapy and 2) after completion of cardiotoxic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female or male with breast cancer tissue diagnosis or a healthy volunteer.
* Plan for treatment as cardiotoxic therapy. Patients for the feasibility study must be post cardiotoxic therapy, and patients for the formal study should not have started the cardiotoxic therapy yet.
* Age ≥ 18 years
* Ability to understand and the willingness to sign a written informed consent
* While all races and ethnicities will be included, subjects must be able to read and speak the English language, and or, the Spanish Language.
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

A female of childbearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

  - Males must be surgically sterile or have a female partner using an acceptable method of contraception.
* Acceptable surgical sterilization techniques are vasectomy with surgery at least 6 months prior to dosing. Males must also refrain from sperm donation during the study and for 6 months following discontinuation of treatment.
* Acceptable methods of contraception for female partners of childbearing potential are an intrauterine device, contraceptive implant, and a barrier method (eg. Condom, diaphragm, cervical cap) during the study and for 6 months after patient discontinuation of treatment.

Exclusion Criteria:

* Patients for the feasibility study must be post cardiotoxic therapy
* Known Type 1 or Type 2 diabetes.
* Subjects who are receiving any other investigational agents that are not compatible with the study.
* Subjects with known remote, macro, metastases will be excluded from this clinical trial because of their poor prognosis.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any contraindication per MRI Screening Form (Appendix A attached) including, but not limited to:

  * Metal Implants and devices contraindicated at 3T.
  * Breast tissue expanders.
  * Non-MR compatible IV port.
  * Claustrophobia.
* Female subjects who are already pregnant.
* Sickle cell disease
* Hemolytic anemia
* If the subject agrees to doing a cardiac function MRI scan with gadolinium based contrast agent intravenously:

eGFR ≤ 30 mL/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Detect subclinical anthracycline induced cardiotoxicity using hyperpolarized carbon-13 pyruvate | 4 years
  Detect the correlation between cardiac carbon-13 pyruvate metabolism and cardiac mechanical function at baseline and after exposure to cardiotoxic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Vlad G Zaha, MD, PhD, Principal Investigator — Advanced Imaging Research Center
Locations (1):
- UT Southwestern - Advanced Imaging Research Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT03685175/ICF_000.pdf